CLINICAL TRIAL: NCT03240198
Title: Marqueurs Biologiques Des Bronchopneumopathies Chroniques Obstructives Professionnelles
Brief Title: Biological Markers for Professional COPD
Acronym: MB2PROF
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Centre Hospitalier Intercommunal Creteil (Other)
Collaborators: Centre Hospitalier Universitaire de Besancon (Other); University Hospital, Bordeaux (Other); University Hospital, Caen (Other); University Hospital, Lille (Other); Centre Hospitalier Le Havre (Unknown); Henri Mondor University Hospital (Other)
Responsible Party: Principal Investigator, Pascal ANDUJAR, Principal Investigator, Centre Hospitalier Intercommunal Creteil
Other Study IDs: MB2PROF
Record Dates: First submitted 2016-09-23; First posted 2017-08-07 (Actual); Last update posted 2017-08-30 (Actual); Status verified 2017-08

CONDITIONS: Copd
Keywords: occupational; cohort; biomarkers
MeSH Terms: conditions — Pulmonary Disease, Chronic Obstructive

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Blood samples
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (2):
- COPD
- Controls

SUMMARY:
Chronic obstructive pulmonary disease (COPD) is a frequent disease, mainly linked to tobacco smoking leading to chronic respiratory failure. It is characterized by an inflammatory spate with modification of protease-antiprotease and oxidant-antioxydant balances. Local modifications are associated with systemic changes. Many occupational factors have been associated with an excess of COPD in epidemiological studies, however without identification of any specific clinical or biological phenotype.

Pathophysiological pathways involved in COPD might be different according to etiologic agents. Therefore, it is important to focus research on blood biomarkers associated with some well-characterized occupational COPD.

The objectives of MB2PROF project are:

1. To build the first multicentric cohort of cases of occupational COPD, with collection of plasma and DNA samples,
2. To study the evolution of clinical and lung function parameters of occupational COPD in comparison with non occupational COPD during a follow-up study,
3. To identify biological phenotypes of COPD associated to a given etiological agent.

The methodology includes:

1. The constitution of a cohort with a clinical and biological follow-up during 5 years. Subjects will be recruited in 7 occupational diseases departments, with the collaboration of Pneumology departments.

   Four groups of males subjects will be recruited (G1 : occupational COPD (6 groups of 60 subjects, corresponding to 6 groups of occupational agents) ; G2 : non occupational COPD (n = 60) ; G3 : subjects with similar occupational exposure to G1 subjects but without COPD (6 groups of 60 subjects) ; G4 : subjects free of occupational exposure and of COPD (n = 60)), paired on tobacco-smoking and age. For each subject, information on clinical data, lung function parameters, occupation history and blood samples will be collected.
2. The identification of biomarkers, using proteomic and genomic approaches according to subgroups (with different etiologies) of occupational COPD,
3. The study of molecular pathways identified in these subgroups, with in vitro and in vivo studies The MB2PROF project is an original and ambitious multidisciplinary and translational project. The constitution of well-characterized COPD cases cohort should allow the identification of biomarkers and molecular pathways associated with some subgroup of subjects, and improve the knowledge of mechanisms involved.

ELIGIBILITY:
Inclusion Criteria:

* COPD

Exclusion Criteria:

* Other obstructive disease

Ages: 40 Years to 80 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: COPD and healthy subjects exposed to tobacco smoking and/or to occupational dust
Sampling Method: Non-Probability Sample
Enrollment: 400 (Estimated)
Dates: Start 2010-01; Primary Completion 2016-01 (Actual); Study Completion 2021-01 (Estimated)

PRIMARY OUTCOMES:
C Protein Reactive | at year 1
blood inflammatory markers | at year 1

SECONDARY OUTCOMES:
C Protein Reactive | every year during 5 years
blood inflammatory markers | every year during 5 years

CONTACTS AND LOCATIONS:
Locations (1):
- CHI Créteil, Créteil, France